CLINICAL TRIAL: NCT00752596
Title: Compassionate Use Study to Assess the Long Term Safety of 125 mg Per Day of Oral Azimilide Dihydrochloride in One Patient Following Termination of the SHIELD Open-label Study 2001060
Brief Title: Compassionate Use Study of 125 mg Per Day of Azimilide Dihydrochloride in One Patient
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Stephen R Marcello, MD, Procter and Gamble Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005076
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Congestive Heart Failure
Keywords: patients; with ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 1 tablet of 125 mg/day of azimilide 2HCl, oral
  Interventions: Drug: Azimilide 2HCl

INTERVENTIONS:
Drug: Azimilide 2HCl — One tablet of 125 mg/day azimilide 2HCl, taken until the study is terminated

SUMMARY:
This is an open-label, long term compassionate use study of 125 mg per day of azimilide 2HCl in a patient who completed two other protocols (2000098 and 2001060.

ELIGIBILITY:
Inclusion Criteria:

* No inclusion criteria as the patient to be included is this compassionate use protocol is currently receiving azimilide therapy

Exclusion Criteria:

* Currently taking Class I or other Class III antiarrhythmic drug or other drugs that may prolong QT interval.
* Is unwilling or unable to give or understand informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
There was no outcome measure in this compassionate use

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marcello, MD, Study Director — Procter and Gamble
Locations (1):
- Research Site, Scottsdale, Arizona, United States